# **Study Title:**

Preventing Alcohol and Other Drug Use and Violence Among Latino Youth

**NCT #:** 

NCT05240313

# **Date of Document:**

June 30, 2021 (original date)

February 10, 2025 (edited for clinicaltrials.gov)

#### **KiR Consent English**

# **Start of Block: Default Question Block**

Q1 **Title of Study:** Preventing Alcohol and Other Drug Use and Violence Among Latinx Youth **CONTACT INFORMATION** 

Principal Investigator: Christopher Salas-Wright, PhD Institution: Boston College School of Social Work

Phone Number: 617-552-1295 Email Address: wrightcu@bc.edu Study Contact Name: J.C. Hodges

Study Contact Phone Number: 617-552-1295 Study Contact Email: hodgesjb@bc.edu

The purpose of this study is to learn how to help Venezuelan youths make good decisions about alcohol, drugs, and violent behaviors. We expect that about 30 youths will be in this research study.

### What Will I be Asked to Do?

If you agree for your child to participate in the study, your child will be asked to do a few things. The first is to take a survey 3 different times.

We will work with your child to schedule a time for the first survey and it will be taken online. The survey will take about half an hour.

Your child will be asked questions about how much they use their phone and the internet, how much they use alcohol, cigarettes, and drugs, and questions about how they feel about different forms of violent behavior. We ask that you give your child privacy to take the survey. Only the researchers will see their answers and they cannot be used against your or your child in any way. Your child will receive \$30 each time he or she complete a survey.

After that, we may ask your child to do two different things. He or she may be asked to participate in weekly sessions for 10 weeks to learn strategies to avoid using alcohol/drugs and aggressive situations. These sessions will be online and have different worksheets, videos, and other ways to help learn. If your child is not asked to participate in the 10 weekly sessions, he or she will be asked to participate in a one-time workshop to learn more about alcohol and drug use and coping skills. He or she will be assigned at random.

Your child will be asked to complete another survey after completing either the 10 week program or the one-time workshop. He or she will be asked to take the survey again after **3** months. Each time he or she will receive another **\$30** dollars.

Your child may also be asked to participate in a focus group (which is a group interview or conversation) after those **3** months. We want to hear about how their experience with the program. Those groups will take about 1-2 hours. We will audio record them so we can write down what everyone says, but the answers will remain confidential and cannot be used against your child. **He or she will receive another \$30 for participating in the focus group.** 

# **Asking for Contact Information**

We will ask you to give us ways to contact you and your child – phone, email, Facebook, Twitter, WhatsApp, et cetera. We are asking for this information so that we can contact you to remind you about the next survey.

What should I think about before I enroll my child in this research?

You should ask any questions you may have and obtain answers before you decide whether to allow your child to be in the study. We want to make sure you get answers to all of your questions. Make sure you ask us any questions you want to. The research study will take about 6 months. Your child may be asked to participate in a ten week program, which is a lot of time!

# Does my child have to be in this research?

No. Your child's participation in this study is voluntary. Your child does not have to be in this study if you do not want to, and he or she can leave the study at any time. Your child will not lose any services, benefits, or rights he or she would normally have if you choose not to have them be in the study or if he or she leaves the study early.

# Is there any way being in this study could be bad for my child?

Taking part in the study involves some small risks. Talking about alcohol, drugs, and violent behavior can be upsetting. We will not ask your child to talk about their own experiences during the program sessions if they don't want – it will be talking about made-up scenarios and practicing different skills. However, if you don't want your child to be in the study, nothing bad will happen to them. If your child becomes upset, you or your child can talk to a counselor on our research team who is a licensed therapist. We will also give you a study phone number to call if you need to talk to someone on the research team and can provide additional resources for other mental health support. Finally, we cannot guarantee anonymity for participating in the focus group as there will be other youth participating. However, we will do everything we can to ensure that confidentiality is maintained by all participants.

# What are the benefits to being in this study?

Your child will learn how to make decisions about difficult topics and communicate those

decisions clearly. If you decide for him or her to be in the study, your child will also help us learn how to help other Venezuelan youths. We are doing this study because we want to learn more about how to help Venezuelan youths make good decisions about alcohol, drugs, and violence and avoid problems. If your child is selected to participate in the ten week program, he or she will also get a t-shirt for their time.

### What happens to the information collected for the research?

We will keep all study records, including recordings and any codes to your data, in a secure location online. Only our research team members will be able to access your data. Passwords will be used to keep people outside our team from seeing your data. Research records will be labeled with a code. A master file that links names and codes will be maintained in a separate and secure location. All electronic files containing identifiable information will be password-protected. Only the members of the research staff will have access to the passwords. At the end of this study, the researchers may publish their findings. Information will be presented in summary format and you will not be identified in any publications or presentations.

Your information may be looked at and/or copied for research or regulatory purposes by:

The National Institutes of Health (NIH); Department of Health and Human Services (DHHS); other government agencies; other Boston College employees for audit and/or monitoring purposes; and other organizations collaborating in the research.

This research is covered by a Certificate of Confidentiality (CoC) from the National Institutes of Health. The researchers with this CoC may not disclose or use information or documents that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding. Your information may not be used as evidence if there is a court subpoena, unless you consent to this use. Information or documents protected by this CoC cannot be disclosed to anyone else who is not connected with the research except as described below, and

If you consent to the disclosure; If it is used for other scientific research as allowed by federal regulations protection research subjects. A Certificate of Confidentiality does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it. If information is revealed that you are at risk to harm yourself or others, to abuse or neglect a child or elderly person, or other forms of abuse, we are required by law to report this immediately to the proper authorities. We will not share any information that you share with your child. We will only share what we are legally required to share.

#### **Payment**

If you agree for your child to participate in this research study, we will give him or her a **\$30** gift card for their time and effort after completing each survey. He or she will also receive a **\$30** gift card for participating in the focus group.

### Who can I talk to?

If you have questions, concerns, or complaints, or think the research has hurt you, talk to Dr. Christopher Salas-Wright at (857) 212-4049 or by email at wrightcu@bc.edu. He speaks both English and Spanish.

This research has been reviewed and approved by an Institutional Review Board ("IRB"). Please contact the director of the Office for Research Protections at Boston College at (617) 552-4778 or irb@bc.edu if:

Your questions, concerns, or complaints are not being answered by the research team.

You cannot reach the research team. You want to talk to someone besides the research team. You have questions about the rights of your child as a research subject. You want to get information or provide input about this research.

### **CONSENT STATEMENT**

I have read this form and the research study has been explained to me. I have been given the chance to ask questions, and my questions have been answered. If I have more questions, I have been told who to call. I agree for my child to be in the research study described above.

I will save or print a copy of this form if I want a copy of it.

Please select one of the following options:

| 0 | Agree for my child to participate (1) | |
|------------|------------------------------------------|-----|
| $\bigcirc$ | Do not agree for my child to participate | (2) |

**End of Block: Default Question Block**